CLINICAL TRIAL: NCT07319117
Title: A Double-blind, Placebo-controlled, Randomised, Acute, Repeated Measures Cross-over Study to Evaluate the Impact of Skoshify 'Think Tank' Nutritional Formulation on Cognitive Performance Following Stress Exposure.
Brief Title: Evaluation of the Impact of a Nutritional Formulation on Cognitive Performance Following Stress Exposure.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Collaborators: Sköshify™ Corporate HQ, 7045 Quiet Retreat Court, Niwot, CO 80503-7174 (Unknown)
Responsible Party: Principal Investigator, Zoe Kolokotroni, Principal Investigator, Leeds Beckett University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P34232
Record Dates: First submitted 2025-12-03; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Assessment; Working Memory; Executive Function (Cognition); Sustained Attention; Inhibitory Control; Cognitive Flexibility; Cortisol; Stress; Anxiety; Depression; Sleep Quality; Blood Pressure; Heart Rate; Mental Fatigue; Physical Fatigue; Productivity; Effort
Keywords: Cognitive Performance; Stress Response; Creatine; Magnesium; L-Tyrosine; L-Theanine; Rhodiola; Phosphatidylserine; Citicoline
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Mental Fatigue; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: This study will follow a double-blind, placebo-controlled, randomised, acute, repeated measures cross-over study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will follow a double-blind, placebo-controlled, randomised, acute, repeated measures cross-over study. Blinding will be maintained for investigators administering the intervention and analysing outcomes. Participants will receive a matched placebo, or active formulation drink matched in appearance, taste and volume. The placebo and active formulations will be administered in a caffeine vehicle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single acute dose (5.6g) of 'Think Tank' Formulation in a caffeine vehicle. (Active Comparator): The active formulation will be dissolved in a 200ml volume coffee beverage (1.8g Nescafe, 50-100mg caffeine). The coffee beverage will be brewed at approximately 90-96◦C. When the beverage has reached a temperature of 65◦C the active nutritional formulation will be added and mixed until dissolved. Each acute dose contains, Magnesium 105mg, Sodium 5mg, Creatine Monohydrate 2.5g, Magnesium Gluconate 2g, L-Tyrosine 500mg, Phosphatidylserine 20% powder 200mg, L-Theanine 200mg, Citicoline Sodium 125mg, Rhodiola Rosea Root Extract 100mg.
  Interventions: Dietary Supplement: Skoshify 'Think Tank' Formulation
- Single acute dose (2.0g) of matched placebo in a caffeine vehicle. (Placebo Comparator): The placebo will be dissolved in a 200ml volume coffee beverage (1.8g Nescafe, 50-100mg caffeine). The coffee beverage will be brewed at approximately 90-96◦C. When the beverage has reached a temperature of 65◦C the placebo will be added and mixed until dissolved. The placebo contains Maltodextrin from corn 1.5mg and Organic acacia gum powder 0.5g.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Skoshify 'Think Tank' Formulation — Each acute dose contains, Magnesium 105mg, Sodium 5mg, Creatine Monohydrate 2.5g, Magnesium Gluconate 2g, L-Tyrosine 500mg, Phosphatidylserine 20% powder 200mg, L-Theanine 200mg, Citicoline Sodium 125mg, Rhodiola Rosea Root Extract 100mg.
  Arms: Single acute dose (5.6g) of 'Think Tank' Formulation in a caffeine vehicle.
Other: Placebo — The placebo contains Maltodextrin from corn 1.5mg and Organic acacia gum powder 0.5g.
  Arms: Single acute dose (2.0g) of matched placebo in a caffeine vehicle.

SUMMARY:
The proposed project will evaluate the synergistic effects of a nutritional formulation, 'Think Tank' on cognitive performance following exposure to a psychological and physical stressor. Adopting a double-blind repeated measures cross-over design, middle-aged females (40-60 years) will be recruited to take part in a two-stage research study that will examine whether the formulation enhances cognitive performance and subjective well-being following the challenge of a stressor, compared to placebo. Cognitive assessments will examine the impact of the nutritional formulation on working memory, sustained attention, cognitive flexibility and inhibitory control. The study will also assess physiological (heart rate, blood pressure and cortisol) and subjective (well-being, anxiety, positive and negative mood, stress) markers of stress reactivity. The study will also explore levels sleep quality, mental and physical fatigue, effort, productivity, and perceived impact of the intervention.

DETAILED DESCRIPTION:
Chronic stress can have a profound impact on quality of life, including cognitive health. Nutritional interventions offer promising, non-pharmacological approaches to support brain health, with particular nutrients showing potential to modulate stress and cognitive function. Creatine, Magnesium, L-Tyrosine, L-Theanine, Rhodiola, Phosphatidylserine and Citicoline have been shown to independently offer cognitive benefits, with the greatest impact observed during episodes of physiological and psychological stress. It is currently unknown whether a combination of these nutrients could produce a synergistic effect on cognitive performance that exceeds the impact of the individual nutrients alone.

This study will follow a double-blind, placebo-controlled, randomised, acute, repeated measures cross-over study design examining cognitive performance, productivity, sleep quality, mental and physical fatigue and subjective/physiological/endocrine responses to an acute psychological and physical stressor following (i) 'nutritional formulation+caffeine' or (ii) 'placebo+caffeine' drink. This research has the potential to identify a novel nutritional intervention that can reduce the negative impacts of stress on cognition.

Participants interested in the study will first take part in an initial health screening to ensure all criteria for eligibility are met. The health screening will include questions on physical and psychological conditions, medication, menstrual cycle, dietary behaviours and supplementation use. Eligible participants will then attend the Human Behavioural Neuroscience Labs at Leeds Beckett University city campus on three occasions over a period of a maximum of 8 weeks.

Prior to all visits participants will be asked to abstain from alcohol and exercise for 24 hours and to fast one hour prior to the session. Participants will also be asked to abstain from caffeine use for a minimum of 6 hours prior to the session. The first visit will involve collection of demographic information and completion of stress, anxiety and depression scales. Daily intake of caffeine consumption and dependency, levels of sleep quality will also be measured. Height and weight will be measured and baseline blood pressure readings taken. Familiarisation with the cognitive tasks will also take place during this visit. Participants will complete the CANTAB battery cognitive tasks to reduce the impact of early practice effects during the test session assessment. Following familiarisation, baseline cognitive performance will also assessed. The CANTAB battery will include the Digit Span (assessment of working memory and attention), Intra-Extra Dimensional Set Shift ( assessment of cognitive shifting and flexibility), Stop-Signal Task (assessment of executive function and inhibitory control) and Rapid Visual Information Processing (assessment of sustained attention).

Experimental test sessions two and three will follow identical procedures. Following a 15-minute resting period, baseline cortisol saliva sample, cardiovascular measures (heart rate and blood pressure), mood state, will be taken. The intervention will then be administered (Formulation + Caffeine) or (Placebo + Caffeine) in 200ml drink and consumed within a 5-minute timeframe. Following a 30 minute absorption period, participants will then be taken to a separate stress-induction room where they will be introduced to the Trier Social Stress Test (TSST). Following completion of the TSST, participants will then complete the Socially evaluated cold pressor test (SECPT). A combination of both the TSST and SCEPT will ensure activation of the both the autonomic and glucocorticoid stress systems and reduce the level of habituation to the stress response across repeated test sessions. The stress protocol will last approximately 20 minutes.

Following stress exposure, the CANTAB battery of cognitive tests will be administered in a serial order. Cognitive assessment will take place during the 40-minute period post-stressor. Throughout the test session cortisol saliva samples, cardiovascular measures (heart rate and blood pressure), mood state, levels of fatigue and perceptions of intervention impact will be measured. Twenty-four hours post session, an online questionnaire assessing the previous night's sleep and levels of productivity since treatment consumption will be administered. Data on side effects and physical experiences following treatment/placebo consumption will also be collected at this time point.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent (in English)
2. Aged 40-60
3. Female
4. Daily caffeine drinkers
5. Healthy and free from significant physical and psychiatric disorders

Exclusion Criteria:

1. Current cigarette smokers/vapers.
2. Known food allergy or intolerance to the investigational products or control products.
3. Not willing to consume coffee.
4. Individuals diagnosed with psychiatric/mental health conditions.
5. Individuals engaging in recreational drug use.
6. Individuals with diagnosed cardiovascular conditions (e.g. heart disease, high blood pressure)
7. Individuals taking prescribed medication except contraceptives/hormone replacement therapy
8. Individuals suffering from Raynaud's or circulatory issues
9. Individuals who have suffered an injury or infection in their hand/arm in the last month
10. Individuals who have suffered from chronic pain conditions or experience extreme numbness or pain in response to cold temperatures.
11. Previous brain injury/brain surgery
12. Individuals who work night shifts.
13. Currently pregnant or breastfeeding.
14. Previous participants in a laboratory stress protocol.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Working Memory Performance | Assessed across 3 timepoints. At baseline (Visit one - Screening) and immediately post stress exposure following consumption of either the active formulation (Visit Two - Test session 1) or placebo (Visit Three - Test session 2).
  Assessed using the Cambridge Neuropsychological Test Automated Battery (CANTAB) Digit Span Task (Forwards and Backwards). The task measures verbal short term working memory. Participants hear a series of digits and are asked to then immediately verbally repeat the sequence, either as it was heard (forwards), or in reverse order (backwards). The forwards tasks assesses verbal working memory and attention, while the backwards span task additionally tests cognitive control and executive function. The primary outcome is the longest sequence problem successfully reached and passed by the subject scored 0 to 9, with a higher score indicating better performance. The total number of attempts made by a subject across all spans reached is also measured, scored 0 to 18, with a lower score indicating better performance.
Cognitive flexibility and attentional set-shifting. | Assessed across 3 timepoints. At baseline (Visit one - Screening) and immediately post stress exposure following consumption of either the active formulation (Visit Two - Test session 1) or placebo (Visit Three - Test session 2)
  Assessed using the Cambridge Neuropsychological Test Automated Battery Intra-Extra Dimensional Set-Shift Task. The task assesses the ability to shift attention between different stimulus dimensions and adapt to changing rules. The outcome measure is the total number of times that the subject chose a wrong stimulus, measured from 0 to 402, and the total number of trials for which the outcome was an incorrect response, measured from 0 to 50. Lower scores indicate better performance.
Sustained attention. | Assessed across 3 timepoints. At baseline (Visit one - Screening) and immediately post stress exposure following consumption of either the active formulation (Visit Two - Test session 1) or placebo (Visit Three - Test session 2)
  Assessed using the Cambridge Neuropsychological Test Automated Battery Rapid Visual Information Processing Task. Participants are presented with digits 2-9 in a pseudo-random order and are requested to detect three -target sequences of digits (e.g. 4-6-8). The primary outcomes are, 'A' the signal detection measure of a subject's sensitivity to the target sequence, scored from 0 to 1 , with higher scores indicating better performance. The RVP Probability of False Alarm, scored 0 to 1 is also measured, with lowers scores indicating a better performance. Median response latency on trials where the subject responded correctly is also calculated.
Inhibitory control | Assessed across 3 timepoints. At baseline (Visit one - Screening) and immediately post stress exposure following consumption of either the active formulation (Visit Two - Test session 1) or placebo (Visit Three - Test session 2)
  Assessed using the Cambridge Neuropsychological Test Automated Battery Stop-Signal Task. The task measures the ability to inhibit a pre-planned, dominant motor response. The main outcome is the Stop Signal Reaction Time, the estimate of time where an individual can successfully inhibit their responses 50% of the time, measured from 0 to 1000, with lower scores indicating better inhibitory control.

SECONDARY OUTCOMES:
Salivary cortisol | Saliva will be collected across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). During each timepoint, a total of 6 samples will be taken during the test session.
  Saliva will be collected via saliva collection aids to assess HPA activity.
Blood pressure | Blood pressure will be measured across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). During each timepoint, a total of 8 blood pressure readings will be taken across the test session.
  Blood pressure will be measured using an ambulatory blood pressure monitor. The blood pressure cuff will be placed on the upper non-dominant arm.
Heart rate | Heart rate will be measured across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). During each timepoint, a total of 8 heart rate epochs readings will be taken across the test session.
  Heart rate will be measured using the H10 Polar heart rate monitor.
Positive and Negative Affect Scale (PANAS) | Assessed across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). At each timepoint the measure will be completed 4 times within the test session, and once four hours post session.
  A 20 item scale assessing two dimensions of positive and negative affect on a 4-point Likert scale from Very slightly/Not at all to Extremely. Scores on each dimension can range from 10 - 50, with higher scores representing higher levels of positive and negative affect.
Visual Analogue Scale (VAS) | Assessed across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). At each timepoint the measure will be completed 7 times within the test session, and once four hours post session.
  A self-devised brief 100mm visual analogue scale assessing dimensions of happiness, sadness, tiredness, anxiety, stress, withdrawal, pain, mental fatigue, physical fatigue, level of focus and effort. Scores range from 0 -100, with higher scores indicating greater levels of each dimension.
Felt Effect Scale | Assessed across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). At each timepoint the measure will be completed 3 times within the test session at 30, 53, ad 95 mins post intervention, and once four hours post session.
  A 6 item VAS assessing perception of intervention impact, measuring items on a 0-100 scale, with higher scores indicating a greater impact.
Leeds Sleep Evaluation Questionnaire | Assessed across 2 timepoints, during Visit Two (Test session 1) and Visit Three (Test session 2). At each timepoint the measure will be completed 2 times, once at the beginning of the test session, and once 24 hours post session.
  a 10-item VAS scale designed to measure changes in subjective sleep quality across areas of getting to sleep, quality of sleep, ease of waking, and early morning behaviour following wakening. Scores range from 0 to 100, with higher scores indicating better sleep quality.
Productivity Scale | Assessed across 2 timepoints (once in each Arm). Assessed once 24 hours post Visit Two (Test session 1) and Visit Three (Test session 2).
  A 5 -item self-devised productivity scale will assess productivity, focus, and mental alertness. Levels of productivity will be assessed via a 0-100 scale, with higher scores indicating greater levels of productivity.
Health Events and Physical Experiences | Assessed across 2 timepoints (once in each Arm). Assessed 24 hours post Visit Two (Test session 1) and Visit Three (Test session 2).
  Participants will be asked to report if they experienced any adverse symptoms in the 24 hours following the test-session, including gastrointestinal symptoms, headaches, dizziness, light-headedness, and mood changes. Participants will be asked to report on the presence and severity of these symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe K Kolokotroni, PhD, Principal Investigator — Leeds Beckett University
Locations (1):
- Leeds Beckett University, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Due to data compliance/ethical restrictions.

REFERENCES:
- [Background] Dassanayake TL, Wijesundara D, Kahathuduwa CN, Weerasinghe VS. Dose-response effect of L-theanine on psychomotor speed, sustained attention, and inhibitory control: a double-blind, placebo-controlled, crossover study. Nutr Neurosci. 2023 Nov;26(11):1138-1146. doi: 10.1080/1028415X.2022.2136884. Epub 2022 Oct 20. PMID 36263942
- [Background] Baba Y, Inagaki S, Nakagawa S, Kaneko T, Kobayashi M, Takihara T. Effects of l-Theanine on Cognitive Function in Middle-Aged and Older Subjects: A Randomized Placebo-Controlled Study. J Med Food. 2021 Apr;24(4):333-341. doi: 10.1089/jmf.2020.4803. Epub 2021 Mar 22. PMID 33751906
- [Background] Magill RA, Waters WF, Bray GA, Volaufova J, Smith SR, Lieberman HR, McNevin N, Ryan DH. Effects of tyrosine, phentermine, caffeine D-amphetamine, and placebo on cognitive and motor performance deficits during sleep deprivation. Nutr Neurosci. 2003 Aug;6(4):237-46. doi: 10.1080/1028415031000120552. PMID 12887140
- [Background] Alvarez XA, Laredo M, Corzo D, Fernandez-Novoa L, Mouzo R, Perea JE, Daniele D, Cacabelos R. Citicoline improves memory performance in elderly subjects. Methods Find Exp Clin Pharmacol. 1997 Apr;19(3):201-10. PMID 9203170
- [Background] Jongkees BJ, Hommel B, Kuhn S, Colzato LS. Effect of tyrosine supplementation on clinical and healthy populations under stress or cognitive demands--A review. J Psychiatr Res. 2015 Nov;70:50-7. doi: 10.1016/j.jpsychires.2015.08.014. Epub 2015 Aug 25. PMID 26424423